CLINICAL TRIAL: NCT01205698
Title: Glycemic Index of Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mead Johnson Nutrition (Industry)
Other Study IDs: 6007
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Glycemic Response

ARMS (4):
- Group 1 - Control A (Placebo Comparator): Vanilla milk-based beverage containing varying levels of lactose, sucrose, and fructose
  Interventions: Other: Nutritional drink
- Group 2 - Experimental A (Experimental): Vanilla milk-based beverage containing varying levels of lactose, sucrose, and fructose
  Interventions: Other: Nutritional drink
- Group 3 - Control B (Placebo Comparator): Vanilla milk-based beverage containing varying levels of lactose, sucrose, and fructose
  Interventions: Other: Nutritional drink
- Group 4 - Experimental B (Experimental): Vanilla milk-based beverage containing varying levels of lactose, sucrose, and fructose
  Interventions: Other: Nutritional drink

INTERVENTIONS:
Other: Nutritional drink

SUMMARY:
This clinical trial will determine the effect of varying types of carbohydrates contained in milk-based beverages on the glycemic response and GI values.

ELIGIBILITY:
Inclusion Criteria:

* male and non-pregnant females 18 - 75 years of age
* signed consent

Exclusion Criteria:

* Known history of chronic illnesses
* Current use of medication or any condition which could make participation dangerous or affect the results
* Unable to comply with experimental procedures
* Food allergies of any kind

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Glycemic Index Laboratories, Toronto, Ontario, Canada